CLINICAL TRIAL: NCT01501370
Title: A Phase II, Multi-center, Open-label, Randomized Study of Vorinostat Plus Lenalidomide and Dexamethasone or Lenalidomide Plus Dexamethasone in Multiple Myeloma Patients Who Experience Biochemical Relapse During Lenalidomide Maintenance Therapy
Brief Title: Vorinostat Plus Lenalidomide and Dexamethasone or Lenalidomide Plus Dexamethasone in Multiple Myeloma Patients Who Experience Biochemical Relapse During Lenalidomide Maintenance Therapy
Acronym: ZLd_Ld
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Tiziana Marangon (Other)
Responsible Party: Sponsor-Investigator, Tiziana Marangon, Sponsor, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNITO-MM-01; 2011-005931-17 (EudraCT Number); RV-MM-PI-0706 (Other: Celgene); MK-0683 -224-00 (Other: MSD)
Record Dates: First submitted 2011-12-16; First posted 2011-12-29 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Biochemical relapse
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Vorinostat; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZLd (Experimental): Patients, who are receiving Lenalidomide maintenance treatment with or without prednisone, will be randomized to receive:
  Cohort 1: ZLd association:
  * Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days
  * Vorinostat orally at the dose of 400 mg/day on days 1-7 and 15- 21 on a 28-day cycle.
  * Dexamethasone orally at the dose of 40 mg day 1,8, 15, 22 every 28 days.
  Interventions: Drug: Vorinostat; Drug: Lenalidomide; Drug: Dexamethasone
- Ld (Active Comparator): Patients, who are receiving Lenalidomide maintenance treatment with or without prednisone, will be randomized to receive: Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days
  • Dexamethasone orally at the dose of 40 mg day 1,8, 15, 22 every 28 days.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Vorinostat — Vorinostat orally at the dose of 400 mg/day on days 1-7 and 15- 21 on a 28-day cycle
  Other Names: Zolinza
  Arms: ZLd
Drug: Lenalidomide — Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days
  Other Names: Revlimid
  Arms: ZLd
Drug: Dexamethasone — Dexamethasone orally at the dose of 40 mg day 1,8, 15, 22 every 28 days.
  Arms: ZLd
Drug: Lenalidomide — Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days
  Other Names: Revlimid
  Arms: Ld
Drug: Dexamethasone — Dexamethasone orally at the dose of 40 mg day 1,8, 15, 22 every 28 days.
  Arms: Ld

SUMMARY:
Histone deacetylase (HDAC) inhibitors represent a potential new class of antitumor agents. Vorinostat (suberoylanilide Hydroxamic acid, SAHA) inhibits the activity of all 11 known human class I and II HDACs. HDACs have many protein targets whose structure and function are altered by acetylation, including histones and non-histones proteins component of transcription factors controlling gene expression and proteins that regulate cell proliferation, migration and death (1). Vorinostat has undergone initial evaluation in several phase I and II clinical trials in both solid and hematologic malignancies. It has shown activity in hematologic malignancies including Hodgkin's disease and non Hodgkin's lymphomas (2-5); it has been approved for treatment of cutaneous manifestation in patients with primary cutaneous T-cell lymphoma who have progressive, persistent or recurrent disease on or following two systemic therapies (6). HDAC function is critical for Multiple Myeloma (MM) cells by actively maintaining a transcriptional program indispensable for their uncontrolled proliferation and/or inappropriate resistance to pro-apoptotic stimuli. The pleiotropic anti-MM effects of Vorinostat and its ability to sensitize MM cellsto multiple conventional or novel agents (7) provide the framework for clinical trials of Vorinostat in MM. A phase I trial of oral Vorinostat alone in advanced MM shows modest activity, but treatment was generally well tolerated (common drug related adverse events (AEs) included fatigue, anorexia, dehydration, diarrhea and nausea and were mostly grade < 2) (8). A phase I clinical trial of Vorinostat in association with Bortezomib in relapsed MM patients report a partial response (PR) rate of 42%, with responses occurring also in patients refractory to a previous Bortezomib based regimen. Treatment was generally well tolerated (main adverse events were myelosuppression, fatigue and diarrhea) (9). Lenalidomide is an active agent against MM, that as shown activity in both the relapse and newly diagnosed settings, in combination with chemotherapy or steroids only. The dose of Lenalidomide commonly used in the relapse setting, in association with steroids, is 25 mg/day on days 1-21 every 28 days (10, 11). A recent phase I study evaluated the safety and tolerability of Vorinostat in combination with Lenalidomide and Dexamethasone in relapsed patients:no dose limiting toxicities prohibited dose escalation, the maximum tolerated dose has not been reached and the maximum administered dose was Lenalidomide 25 mg/day on days 1-21, Dexamethasone 40 mg/day on days 1,8,15,22, Vorinostat 400 mg/day on days 1-7 and 15-21; each cycle was repeated every 28 days. Rate of at least PR was 51%, and activity was seen also in patients who received prior Lenalidomide therapy (clinical benefit reported in 69% of patients, including minimal response or better in 33% of Lenalidomide refractory patients). The most common drug related grade > 3 AEs were neutropenia, thrombocytopenia, diarrhea, anemia and fatigue (12). Since Vorinostat has shown efficacy also in patients previously treated with Lenalidomide, and in patients refractory to Lenalidomide, the investigators hypothesis is that the addition of Vorinostat and low-dose dexamethasone to Lenalidomide (ZLd), in patients experiencing a biochemical relapse during a Lenalidomide maintenance ongoing therapy, can overcome Lenalidomide-drug resistance and result in a significant response rate, that can translate into a significant improvement in survival of MM patients. The second hypothesis is that, since the dose of Lenalidomide commonly administered in maintenance therapy, is 10 mg days 1-21 every 28 days, the increase in Lenalidomide dose to the standard dose used for relapsing patients, plus low-dose Dexamethasone (Ld), in patients experiencing a biochemical relapse during a Lenalidomide ongoing maintenance, can as well overcome Lenalidomide-drug resistance and determine a significant response rate, that can translate into a significant improvement in survival of MM patients.

This is a multicenter non comparative, randomized, open label, phase II study. Patients, who are receiving Lenalidomide maintenance treatment with or without prednisone, will be randomized to receive:

Cohort 1: ZLd association:

Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days Vorinostat orally at the dose of 400 mg/day on days 1-7 and 15- 21 on a 28-day cycle.

Dexamethasone orally at the dose of 40 mg day 1,8, 15, 22 every 28 days.

Cohort 2: Ld association:

Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days Dexamethasone orally at the dose of 40 mg day 1,8, 15, 22 every 28 days.

Patients must have a -confirmed diagnosis of relapsed multiple myeloma. In this Phase II study, a total of up to 35 patients in the ZLd cohort and 48 in the Ld cohort will be enrolled. It is anticipated that full accrual to this study will take approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal for 24 consecutive months or surgically sterilized or agree to continuous abstinence from heterosexual sexual contact or willing to use effective contraception for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of therapy; female patients not pregnant or nursing; female with a negative pregnancy test.
* Male patient agrees to use an acceptable method for contraception during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of therapy.
* Patient diagnosed with MM based on standard criteria, and has measurable disease (14,15), defined as follows:
* Secretory myeloma: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein), and/or where applicable, urine light-chain excretion of > 200 mg/24 hours or involved free light chain (FLC) level > 10 mg/dl provided serum FLC ratio is abnormal;
* Non-secretory myeloma: > 30% plasma cells in the bone marrow and at least one plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e., MRI or CT scan).
* Patient receiving Lenalidomide maintenance therapy as part of first line treatment (concomitant use of prednisone is accepted) and has experienced a biochemical relapse, with evidence of progressive disease defined as increase of 25% from lowest response value in any one or more of the following: Serum M-component (absolute increase must be ≥ 0.5 g/100 ml) and/or Urine M-component (absolute increase must be ≥ 200 mg per 24 h); only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/l) (12).
* No evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically hypercalcemia (serum calcium ≥ 11.5 mg/100 ml) or renal insufficiency (serum creatinine > 1.73 mmol/l), or anemia (hemoglobin value of > 2 g/100 ml below the lower limit of normal or a hemoglobin value < 10 g/100 ml) or bone lesions (lytic lesions, severe osteopenia or pathologic fractures) (11).
* Patient has a Karnofsky performance status ≥ 60%.
* Patient has a life-expectancy > 3 months.
* Patient has not active infectious hepatitis type B or C and no known HIV infection.
* Patient has not to have congenital long QT syndrome or right bundle branch block + left anterior hemiblock (bifascicular block).

Screening ECG with a QTc < 450 msec.

* Patient has not to take anti-arrhythmic drugs or other medicinal products which led to QT prolongation and cumulative high dose of anthracycline.
* Patient has not clinically significant illness that would, in the investigator's opinion, increase the patient's risk for toxicity.
* Patient has not a currently active malignancy, other than non melanoma skin cancer and carcinoma in situ of the cervix. Patients are not considered to have a currently active second malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years and are considered by their physicians to be at less than 30% risk of relapse.
* No history of allergic reactions attributed to study agents.
* No prior exposure to HDACi. Patients exposed to valproic acid could be eligible with a wash out period of at least 30 days.
* More than 30 days since prior class Ia, Ib and Ic antiarrhythmic medications.
* Patient has the following laboratory values within 28 days before baseline day 1 of the cycle 1:
* Platelets count ≥ 75 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
* Aspartate transaminase (AST), Alanine transaminase (ALT), total bilirubin: ≤ 2 x the upper limit of normal (ULN).
* Calculated or measured creatinine clearance: ≥ 20 mL/minute
* PT and PTT: ≤ 1.5 the ULN
* Serum potassium ≥ LLN
* Serum magnesium ≥ LLN
* Serum phosphorus ≥ LLN

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness or social situation that would prevent the subject from signing the informed consent form or limit the compliance with study medications and requirements.
* Pregnant or beast feeding females.
* Use of any other concomitant standard/experimental anti-myeloma drug or therapy.
* Known positive for HIV or active infectious hepatitis, type B or C.
* Known congenital long QT syndrome or right bundle branch block + left anterior hemiblock (bifascicular block).
* Screening ECG with a QTc > 450 msec.
* Ongoing therapy with anti-arrhythmic drugs or other medicinal products which led to QT prolongation and cumulative high dose of anthracycline.
* Patient with currently active malignancy, other than non melanoma skin cancer and carcinoma in situ of the cervix. Patients are not considered to have a currently active second malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years and are considered by their physicians to be at less then 30% risk of relapse.
* History of allergic reactions attributed to study agents.
* Prior exposure to HDACi. Patients exposed to valproic acid could be eligible with a wash out period of at least 30 days.
* Less than 30 days since prior class Ia, Ib and Ic antiarrhythmic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Rate of PR (PARTIAL RESPONSE) with the association of ZLd and Ld | Responses will be evaluated after 112 days from enrollment of each patients (4 cycles of therapy)
  Determine the rate of PR with the association of ZLd and Ld in patients who experience biochemical relapse during Lenalidomide maintenance therapy. ZLd and Ld: responses will be evaluated after the enrollment of 10 and 18 pts respectively. If ≤1 and ≤2 respectively responses will be observed the trial will be stopped. Otherwise 19 and 25 pts respectively will be enrolled: if ≤5 for Zld and ≤7 for Ld responses will be observed, no further investigation will be needed

SECONDARY OUTCOMES:
duration of progression free survival | date of randomization to date of first documentation of progression from any cause, assessed every 3 months from removal of treatment, for approximately 2 years
  The occurrence of progression will determine the duration of PFS.
Overall survival | date of randomization to date of death from any cause, assessed every 3 months from removal of treatment, for approximately 2 years
  The occurence of death will determine the OS

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Palumbo, MD, Principal Investigator — Division of Hematology, University of Turin, Italy
Locations (8):
- Italy (8):
  - Clinica di Ematologia, A.O.U. Ospedali Riuniti, Ospedale Umberto I di Ancona, Ancona, Ancona
  - U.O.S. di Ematologia, Ospedale Mazzoni, Ascoli Piceno, Ascoli Piceno
  - Dh ematologia, A.O.U. Careggi, Florence, Firenze
  - Ematologia, Ospedale S. Maria della Misericordia, Perugia, Perugia
  - Ematologia e Immunoematologia, Azienda Ospedaliera Riuniti Marche Nord, Pesaro, Pesaro
  - Dip. Ematologia-U.O di Ematologia Generale-Azienda USL di Pescara-P.O. dello Spirito Santo, Pescara, Pescara
  - Ematologia , A.O.U. Pisana, Pisa, Pisa
  - Universitaria di Ematologia, A.O.U. San Giovanni Battista di Torino,, Torino, Torino